CLINICAL TRIAL: NCT03108625
Title: Long-term, Open-label, Flexible-dose, Continuation Extension Study With Vortioxetine in Child and Adolescent Patients With Major Depressive Disorder (MDD) From 7 to 17 Years of Age
Brief Title: Continuation With Vortioxetine in Child and Adolescent Patients With Major Depressive Disorder (MDD) From 7 to 17 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12712B; 2015-002658-11 (EudraCT Number)
Record Dates: First submitted 2017-03-10; First posted 2017-04-11 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Depressive Disorder, Major
Keywords: children; adolescent
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vortioxetine (Experimental): Once daily dosing of vortioxetine (oral tablets) for 78 weeks.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Target dose is 10 mg/day; the dose can be down- or uptitrated to 5, 15, or 20 mg/day.
  Other Names: Brintellix; Lu AA21004

SUMMARY:
Evaluation of the long-term safety and tolerability of vortioxetine in child and adolescent patients with a Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5™) diagnosis of MDD

ELIGIBILITY:
Inclusion Criteria:

* The patient is a male or female child aged ≥7 and <12 years or an adolescent aged ≥12 and ≤17 years at Baseline in Study 12712B.
* The patient must have completed extension Study 12712A immediately prior to enrolment into this extension study.
* The patient had a primary diagnosis of a MDD at entry in Study 12709A or 12710A, diagnosed according to DSM-5™.
* The patient is still indicated for long-term treatment with vortioxetine according to the clinical opinion of the investigator.

Exclusion Criteria:

* The patient has been diagnosed with another psychiatric disorder (for example mania, bipolar disorder, schizophrenia or any psychotic disorder) during study 12712A.
* The patient has an attention-deficit/hyperactivity disorder (ADHD) that requires a pharmacological treatment other than a stimulant medication.

Other protocol-defined inclusion and exclusion criteria may apply

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety) | Up to Week 104
  Based on safety assessments (e.g. paediatric adverse event rating scale (PAERS), clinical safety laboratory tests (including reproductive hormones), vital signs, weight, height, Tanner score, menstrual cycle, ECG, and C-SSRS

SECONDARY OUTCOMES:
Change in CDRS-R total score | Change from study 12712A baseline to Week 104
  Children Depression Rating Scale, revised version
Number of relapses (CDRS-R ≥40 with a history of 2 weeks of clinical deterioration) | Up to Week 104
  Number of relapses (CDRS-R ≥40 with a history of 2 weeks of clinical deterioration)
Loss of remission (CDRS-R <28 with a history of 2 weeks of clinical deterioration) | Up to Week 104
  Loss of remission (CDRS-R <28 with a history of 2 weeks of clinical deterioration)
Change in CGI-S score | Change from study 12712A baseline to Week 104
  Clinical Global Impression - Severity of Illness
CGI-I score | Week 104
  Clinical Global Impression - Global Improvement
Children (7-11 years): change in BRIEF using the Global Executive Composite score | Change from study 12712A baseline to Week 104
  Behaviour Rating Inventory of Executive Function
Children (7-11 years): change in BRIEF using the Megacognition Index | Change from study 12712A baseline to Week 104
  Behaviour Rating Inventory of Executive Function
Adolescents (12-17 years): change in BRIEF-SR using the Global Executive Composite score | Change from study 12712A baseline to Week 104
  Behaviour Rating Inventory of Executive Function, Self-report version
Adolescents (12-17 years): change in BRIEF-SR using the Megacognition Index | Change from study 12712A baseline to Week 104
  Behaviour Rating Inventory of Executive Function, Self-report version
Change in CGAS score | Change from study 12712A baseline to Week 104
  Children's Global Assessment Scale
Change in PedsQL VAS score | Change from study 12712A baseline to Week 104
  Pediatric Quality of Life Inventory Present Functioning Visual Analogue Scales

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (31):
- Bulgaria (2):
  - MHAT "Targovishte" AD, Targovishte
  - DCC Mladost-M, Varna
- Marienthal Center of Psychiatry and Psychology, Tallinn, Estonia
- CHU de Nantes - Hopital Hotel Dieu, Nantes, France
- Rheinhessen-Fachklinik Mainz, Kinder und Jugendpsychiatri, Mainz, Germany
- Hungary (2):
  - Vadaskert Alapitvany, Budapest
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza, Gyula
- Italy (2):
  - Scientific Institute Fondazione Stella Maris, Calambrone
  - Universita degli Studi di Messina - Facolta di Medicina e Chirurgia, Messina
- Linda Keruze's Psychiatric Center, LLC, Liepāja, Latvia
- Poland (6):
  - Prywatne Gabinety Lekarskie ¿Promedicus¿ Anna Agnieszka Tomczak, Bialystok
  - Centrum Badan Klinicznych PI-House Sp. z o.o., Gdansk
  - Przychodnia Syntonia Poradnia Zdrowia Psychicznego, Kielce
  - SPECTRUM Centrum Neurologii i Psychiatrii, Lublin
  - Filip Rybakowski Specjalistyczna Praktyka Lekarska, Poznan
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej (SPZOZ) - Centrum Neuropsychiatrii "NEUROMED", Wroclaw
- Russia (9):
  - Specialized Clinical Psychiatric Hospital 1 of the Ministry of Health, Krasnodar
  - Lipetsk Regional Psychoneurological Hospital, Lipetsk
  - Nizhny Novgorod Region State Institution Of Healthcare, Nizhny Novgorod
  - Medicorehabilitation Research Center "Phoenix", Rostov-on-Don
  - Rostov State Medical University of the Minzdravsotsrazvitiya of Russia, Rostov-on-Don
  - Guz "Saratov Regional Psychiatric Hospital St. Sofii", Saratov
  - Saratov State Medical University, Saratov
  - State Budgetary Healthcare Institution, Tonnel’nyy
  - State Budgetary Healthcare Institution of Sverdlovsk Region, Yekaterinburg
- Serbia (2):
  - Clinic of Neurology and Psychiatry for Children and Adolescents, Belgrade
  - Clinical Center of Vojvodina - Clinic of Psychiatry, Novi Sad
- Cape Trial Centre, Bellville, South Africa
- Spain (2):
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Unidad de Salud Mental Infanto-Juvenil (USMI-J) Edificio de Consultas Externas. Hospital MarAtimo, Torremolinos
- Alder Hey Childrens Hospital, Liverpool, United Kingdom